CLINICAL TRIAL: NCT06309979
Title: A Multicenter, Observational Study to Characterize Growth in Children With Idiopathic Short Stature
Brief Title: A Study to Assess Growth in Children With Idiopathic Short Stature
Status: Recruiting | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 111-903
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Short Stature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study 111-903 will generate baseline growth data in children with ISS by collecting growth measurements and other variables of interest.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be > 2 years old, and ≤ 14 years old (female) or ≤ 16 years old (males) at the time of signing the informed consent.
2. A height assessment corresponding to a height Z-score of ≤ -2.25 SDs in reference to the general population of the same age and sex, as calculated using the Centers for Disease Control and Prevention (CDC) growth chart (https://www.cdc.gov/growthcharts/zscore.htm).
3. Participants who have either never received hGH, or who are currently receiving hGH treatment.
4. Historic stimulation test result with serum or plasma GH level greater than 10 μg/L.
5. Parent(s) or guardian(s) are willing and able to provide written, signed informed consent.

Exclusion Criteria:

1. Diagnosis of systemic disease or condition that may cause short stature, eg renal, neoplastic, pulmonary, cardiac, gastrointestinal, immunologic and metabolic disease. Children with such diagnoses can be considered for inclusion if their condition is well controlled, at the discretion of the Medical Monitor.
2. Known presence of one or more pituitary hormone deficiencies
3. Bone age advanced over chronological age by more than 3 years.
4. For hGH naïve participants, historic stimulation test result with serum or plasma GH level greater than 10 μg/L or serum IGF-1 in the normal range for age (between -1.00 SDs and +2.00 SDs).
5. For participants currently on hGH treatment, historic results before GH treatment of stimulation test with serum or plasma GH level greater than 10 μg/L or serum IGF-1 test between -1.00 SDs and +2.00 SDs.
6. Have received an investigational product (IP) or investigational medical device for any purpose within 6 months before the Screening visit. .

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include up to 600 pediatric individuals with Idiopathic Short Stature.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in annualized growth velocity (AGV) | Every 6 months through end of study, up to 15 years
Change in Height Z-score | Every 6 months through end of study, up to 15 years
Change in Standing Height | Every 6 months through end of study, up to 15 years
Change in BMI | Every 6 months through end of study, up to 15 years
Change in BMI Z-score | Every 6 months through end of study, up to 15 years

SECONDARY OUTCOMES:
Frequency of event rates of medical events of interest | Every 6 months through end of study, up to 15 years
Frequency of Serious Medical Events | Every 6 months through end of study, up to 15 years
Association between specific variants and growth velocity | Every 6 months through end of study, up to 15 years
Association between other health outcomes directly related to short stature | Every 6 months through end of study, up to 15 years

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Phoenix Children's Hospital - Thomas Campus (Main), Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Harbor-UCLA Medical Center - The Lundquist Institute (Los Angeles Biomedical Research Institute (LA BioMed), Los Angeles, California
  - Children's Hospital of Orange County Main Campus - Orange, Orange, California
  - Center Of Excellence in Diabetes and Endocrinology, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - Children's National Health System, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Health System - Corporate Headquarters, Pensacola, Florida
  - Centricity Research, Columbus, Georgia
  - St. Luke's Children's Endocrinology, Boise, Idaho
  - Rocky Mountain Diabetes Center - Idaho Falls, Idaho Falls, Idaho
  - Rocky Mountain Clinical Research - Idaho Falls, Idaho Falls, Idaho
  - University of Louisville School Of Medicine - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner Health Center for Children - New Orleans, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Medical School - Masonic Children's Hospital - Pediatric Specialty Care Explorer Clinic, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Iowa Stead Family Children's Hospital, Princeton, New Jersey
  - UBMD Pediatrics, Buffalo, New York
  - ACGC Research, NYU Ambulatory Care Garden City, Garden City, New York
  - New York University Grossman School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai (ISMMS) - The Mount Sinai Hospital (MSH) - Pediatric Associates, New York, New York
  - Montefiore Medical Center (MMC) - The Children's Hospital at Montefiore (CHAM), The Bronx, New York
  - WakeMed Children's - Pediatric Endocrinology - North Raleigh, Raleigh, North Carolina
  - Cincinnati Children's Hospital Medical Center Burnet Campus, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Prisma Health Children's Hospital - Midlands, Columbia, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Endocrinology, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Charleston Area Medical Center (CAMC) Health System, Charleston, West Virginia
  - Medical College of Wisconsin, Children's Hospital, Milwaukee, Wisconsin